CLINICAL TRIAL: NCT05849857
Title: Phase II Multicenter Clinical Trial: Mosunetuzumab for Early Relapse of Follicular Lymphoma in the Nordic Countries
Brief Title: Mosunetuzumab for Early Relapse of Follicular Lymphoma in the Nordic Countries
Acronym: MERLIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Hoffmann-La Roche (Industry); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Brodtkorb, Senior consultant, Department of Oncology, Principal Investigator, M.D., Ph.D., Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU CT NO: 2022-500100-21-01; NLG-FL6 (Other: The Nordic Lymphoma Group); ML43841 (Other: Roche)
Record Dates: First submitted 2023-03-22; First posted 2023-05-09 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Phase II, one arm, open label clinical trial of subcutaneous mosunetuzumab mono-therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subcutaneous mosunetuzumab (Experimental): The duration of each treatment cycle is 21 days.
  Cycle 1 Day 1:
  5 mg Mosunetuzumab SC
  Cycle 1 Day 8:
  45 mg Mosunetuzumab SC
  Cycle 1 Day 15:
  45 mg Mosunetuzumab SC
  Cycle 2-8 Day 1:
  45 mg Mosunetuzumab SC
  Patients in complete remission after 8 cycles enter follow-up. Patients with stable disease or partial remission can receive up to a total of 17 cycles:
  Cycle 9-17 Day 1:
  45 mg Mosunetuzumab SC
  Interventions: Drug: Mosunetuzumab

INTERVENTIONS:
Drug: Mosunetuzumab — Mosunetuzumab is administered as a subcutaneous injection. The first dose is 5 mg in 0,5 mL volume, subsequent doses are 45 mg in 1,0 mL volume.
  Other Names: Dexamethasone

SUMMARY:
In this clinical trial adult patients diagnosed with follicular lymphoma and relapse or progression of disease within 24 months of starting first line treatment will be treated with mosunetuzumab. This is a bispecific antibody, a new type of immunotherapy that redirects the bodies own immune cells (T-cells) to attack and kill the lymphoma cells. The main question the trial aims to answer is if mosunetuzumab works better than standard treatments in this sub-group of patients. Patients will receive mosunetuzumab as injections in the abdominal subcutaneous fat once a week for the three first doses, then every third week 7 times. If all signs of disease are gone as evaluated by PET-CT images, the treatment is stopped. If signs of disease remain on PET-CT images, the patients can receive treatment every third week for up to a total of one year. After the end of treatment, patients are followed two years in the trial for signs of progression or relapse.

DETAILED DESCRIPTION:
Background: Standard first line treatment for patients with follicular lymphoma and symptomatic disease is immunotherapy with or without chemotherapy. The most commonly used treatment regimens are rituximab plus bendamustin or CHOP (cyclophosphamide, doxorubicin, vincristine and prednisolone), rituximab plus lenalidomide or rituximab monotherapy. The long-term outcome is similar for these regimens; 75-80% of patients are alive 10 years after initial treatment. A subgroup of 20-40% of patients does not respond to or relapse within 24 months of initial treatment (abbreviated POD24 for "progression of disease within 24 months), and they risk poorer effect of second line treatments and shorter survival. Only 30-70% of these patients are alive 5 years after initial treatment, depending on the type of first line treatment, and they are in need of improved treatment options. Mosunetuzumab is a new, bispecific, T-cell engaging antibody that has shown very high response rates and long response duration in B-cell lymphoma patients with multiple relapses or lack of response to standard salvage regimens. It is therefore possible that mosunetuzumab will benefit patients with POD24. The main hypothesis of this trial is that mosunetuzumab is better than standard 2nd line salvage regimens in terms of progression free survival 2 years after the initiation of 2nd line treatment in POD24 patients.

Objectives: The main objective is to investigate the efficacy of subcutaneous (SC) mosunetuzumab monotherapy in follicular lymphoma (FL) with POD24.

The secondary objectives are to investigate

* safety of mosunetuzumab in patients with a current POD24 event
* prognostic significance of 18F-FDG-PET-CT response to mosunetuzumab
* rate of transformation to higher grade lymphoma following mosunetuzumab
* patients´ self-reported quality of life during and after mosunetuzumab
* resource usage related to mosunetuzumab

Interventions: Mosunetuzumab is administered SC as described below. Patients are followed for at least 2,5 years and a maximum of 5 years in the trial. Study-specific sampling of peripheral blood for exploratory research amounts to 330-380 mL (depending on the number of treatment cycles) collected over 3 years. Study-specific tumor samples for future research will be collected by fine needle aspiration before the start of treatment and after the third treatment cycle.

Ethical considerations: Previous studies have shown that mosunetuzumab is highly effective and well tolerated in heavily treated B-cell lymphoma patients. The safety profile is favourable compared to standard immunochemotherapy. Mosunetuzumab can be safely administered to older patients with co-morbidities, and there is no upper age limit for participation in the trial. The potential beneficial effect of mosunetuzumab in a population of follicular lymphoma patients with POD24 outweighs the risk for rare and undiscovered serious adverse events. The total volume of blood samples is considered acceptable for patients in clinical trials. The extra tumor samples for research purposes will only be collected if deemed safe and not to cause unreasonable discomfort for the participating subject. The extra number of CT scans is 2-3 compared to standard practice and represents a minimal increase in radiation exposure. In total, the benefit to risk balance is deemed positive for this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent according to ICH-GCP guidelines.
2. Age ≥ 18 years.
3. Follicular lymphoma grade 1-3a with a current relapse or progression within 24 months of starting 1st line treatment or refractory to 1st line treatment (POD24), more specifically:

   1. Documented current relapse or progression of FL within 24 months of starting first line treatment containing a monospecific anti-CD20 antibody (such as rituximab or obinutuzumab with or without chemotherapy, small molecular inhibitors or immunomodulating agents such as lenalidomide).
   2. Current lack of response/refractoriness to first line treatment, i.e., no objective response or documented progression within 6 months following at least four cycles of monotherapy with a monospecific anti-CD20 antibody (such as rituximab 375mg/m2 iv or 1400 mg SC or equal) or following at least three cycles of a monospecific anti CD20 antibody combined with chemotherapy, small molecular inhibitors or immunomodulating agents such as lenalidomide.
   3. Received one prior treatment line of systemic therapy.
   4. Patients may have had a period of watch and wait before the initiation of first line treatment.
   5. Patients may have received localized radiotherapy previously.
4. At least one two-dimensionally measurable lesion with a longest diameter >15mm.
5. WHO performance status 0-2. Patients with reduced WHO performance status (> 2) can be considered if reduction in performance is caused by the lymphoma as determined by the investigator.

Exclusion Criteria:

1. Received 2 or more previous treatment lines.
2. Grade 3b FL.
3. CD20-negative lymphoma.
4. CNS involvement (current or previous).
5. Impaired bone marrow function (neutrophils < 1.0 x 109/L or platelets < 50 x 109/L) unless due to lymphoma involvement.
6. Severe cardiac disease: impaired cardiac function (NYHA class III or IV), myocardial infarction within the last 6 months, unstable arrythmias and/or unstable angina pectoris.
7. Impaired liver function not caused by lymphoma, defined as serum total bilirubin ≥ 1.5 x ULN (unless elevated due to Gilbert's syndrome) or serum ALT and AST > 3 x ULN.
8. Impaired renal function not caused by lymphoma, defined as calculated creatinine clearance ≤ 40 ml/minute.
9. Other major organ dysfunction not caused by lymphoma.
10. Known history of drug induced liver injury, chronic active hepatitis C (HCV), chronic active hepatitis B (HBV), alcoholic liver disease, primary biliary cirrhosis, on-going extra-hepatic obstruction caused by cholelithiasis, cirrhosis of the liver or portal hypertension.
11. Active severe infection.
12. Hepatitis B (HBV) or hepatitis C (HCV) infection: Subjects with a previous hepatitis B infection will be eligible if they are negative for HBV-DNA; these subjects must be given prophylactic antiviral therapy. Subjects with a previous HCV infection will be eligible if they are negative for HCV-RNA.
13. Known or suspected chronic active Epstein-Barr virus (EBV) infection.
14. Received systemic immunosuppressive medications (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within two weeks prior to the first dose of mosunetuzumab.
15. Administration of live vaccines within four weeks of the first dose of mosunetuzumab or anticipation that live vaccine will be required during the study.
16. History of severe allergic or anaphylactic reactions to chimeric, human, or humanized antibodies, or fusion proteins.
17. Known or suspected hemophagocytic syndrome.
18. Prior allogeneic hematopoietic stem cell transplant.
19. Other current severe medical problems or expected survival of less than approximately five years for non-lymphoma reasons.
20. Current or previous other malignancy within three years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other non-invasive or indolent malignancy without sponsor approval.
21. Psychiatric disorder or dementia which make the patient unable to give an informed consent and/or adhere to the schedule.
22. Pregnancy or breast-feeding.
23. HIV positivity: Subjects that are on HIV-treatment with undetectable HIV-RNA and CD4-counts above 200 will be eligible.
24. Women of reproductive potential not agreeing to use an acceptable method of birth control during treatment and for three months after completion of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
PFS | From the date of starting treatment to the date of first documented progression of disease or death of any cause, whichever came first. Patients will be observed for a minimum of 2 years and a maximum of 4 years for the primary outcome
  Progression free survival

SECONDARY OUTCOMES:
ORR | At the end of 8 cycles (each cycle is 21 days)
  Overall response rate assessed by PET-CT
CRR | At the end of 8 cycles (each cycle is 21 days)
  Complete response rate assessed by PET-CT
DOR | From the date of first documented response to the date of first documented disease progression or death from any cause. Patients will be observed for a minimum of 2.5 years and a maximum of 5 years for the DOR
  Duration of response
TTNT | From the date of starting study treatment to the date of starting 3rd line therapy due to progression of disease or to death of any cause, whichever came first. Patients will be observed for a minimum of 2.5 years and a maximum of 5 years for TTNT.
  Time to new lymphoma treatment
OS | From the date of inclusion to the date of death of any cause. Patients will be observed for a minimum of 2.5 years and a maximum of 5 years for OS.
  Overall survival
The percentage of patients with adverse events | From inclusion until 30 days after last dose of study drug
  Safety and tolerability
The percentage of patients with transformation to aggressive lymphoma | From inclusion to the end of follow-up. Patients will be observed for a minimum of 2.5 years and a maximum fo 5 years.
  The rate of higher grade lymphoma transformation

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Brodtkorb, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (3):
- Helsinki University Hospital, Helsinki, Finland
- Norway (2):
  - Oslo University Hospital, Oslo
  - St. Olavs hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No
Individual participation data will not be shared